CLINICAL TRIAL: NCT04574609
Title: Evaluation of the Impact of the Use of Hypnotherapy Performed by a Virtual Reality Tool Along the Care Pathway of Patients Undergoing Breast Cancer Treatment: Randomized Controlled Trial.
Brief Title: Evaluation of the Impact of the Use of Hypnotherapy Performed by a Virtual Reality Toolalong the Care Pathway of Patients Undergoing Breast Cancer Treatment.
Acronym: HYGEE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HYGEE
Record Dates: First submitted 2020-09-10; First posted 2020-10-05 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: hypnotherapy; virtual reality; anxiety; pain
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no hypnotherapy (No Intervention): A "control" group of patients receiving the usual management for PAC and chemotherapy sessions.
- hypnotherapy (Experimental): A "hypnotherapy" group of patients benefiting from hypnotherapy sessions prior to PAC and chemotherapy cures in addition to the usual management.
  Interventions: Device: Oncomfort® clinical virtual reality

INTERVENTIONS:
Device: Oncomfort® clinical virtual reality — hypnotherapy" arm, patients will receive in addition to the care provided by the usual :
  * for PAC insertion: a 45-minute hypnotherapy session 2 hours before the procedure in a room of the outpatient surgery unit (UCA).
  * during the entire duration of chemotherapy (and/or immunotherapy for HER2+ patients) : one hypnotherapy session before the first treatment and then every 3 weeks. One hypnotherapy session before the first treatment and then every 3 weeks. Thus, sessions will take place before each treatment for 3-week inter-course regimens and every 3 treatments for chemotherapy administered on a weekly. Each session will last 20 minutes.
  Arms: hypnotherapy

SUMMARY:
In 2017, it is estimated that nearly 60,000 new cases of breast cancer will be diagnosed in France. Although several treatments are indicated in this context, chemotherapy remains a curability option whose place today extends to small tumors to support its increasingly approved administration contributing to a continuous increase in survival rates.

However, diagnostic procedures and anti-cancer treatments are frequently responsible for toxicity that can reach high levels of severity and even generate sequelae.

These physical and psychological after-effects of breast cancer treatment have a short and medium-term impact on the quality of life of the patients treated: anxiety, fear, pain, job loss, and the onset of precariousness.

In addition, surgical procedures such as PAC and pic-line surgery are often associated with anxiety and pain. Chemotherapy is particularly associated with anxiety, stress, fatigue, nausea and vomiting.

Some immediate, delayed or even anticipated side effects are not always effectively controlled by the medication available to us. Anti-nausea medications can lead to drug interactions and/or other adverse effects. The interest of a non-drug approach is to get rid of these adverse effects. However, it is underestimated and therefore currently not integrated into current practice.

Its benefits must therefore be explored within the framework of in-depth research protocols that justify our study.

DETAILED DESCRIPTION:
The use of virtual reality (VR) technology as a non-pharmacological tool has developed public interest in improving the control of certain adverse effects induced by chemotherapy. A few small studies suggest that the use of VR during chemotherapy helps reduce anxiety, fatigue and nausea and vomiting. Schneider showed improvement in stress-related symptoms such as anxiety in children aged 10 years and older receiving chemotherapy treatment during a VR session.

A similar study showed a reduction in anxiety in patients receiving chemotherapy for breast cancer treatment coupled with VR. Dr. Hoffman is recognized as a pioneer in the use of VR, which he has proven to be effective in the care of burn patients, coupled with a technique that some have called VR analgesia. He has demonstrated that this technology used in this setting is a novel non-pharmacological approach to improving pain control.

Our project involves the use of a VR module associated with an application delivering hypnotherapy combined with cognitive behavioral therapy that could help improve the adverse effects attributable to chemotherapy. The hypnotherapy that has been shown to be medically effective since its discovery by Mesmer is Ericksonian hypnosis. It usually involves an exchange between the therapist and the patient over a period of time.

marked (suggestion, induction, fascination, dissociation, amplification) which has evolved in our institution in a less elaborate form called "conversational hypnosis".

In this context, VR hypnotherapy appears to be a promising alternative. To date, there are a few studies that demonstrate the reduction of anxiety through the use of this tool during the application of PACs and pick-lines.

The innovation of this study is to report the effects of a combination of hypnotherapy using VR through a program aimed at modifying the experience of adverse effects due to PAC and chemotherapy in the care pathway of breast cancer patients.

It will also be compared to what is called in our institution and practiced routinely: conversational hypnosis which is not Ericksonian hypnosis strictly speaking but because of the parameters mentioned above: time, human resources load has become a simple benevolent conversation that welcomes the patient in every step of his care.

ELIGIBILITY:
Inclusion Criteria:

* Woman whose age ≥ 18 years old
* Negative pregnancy test for women of childbearing age
* Francophone patient
* Patient newly diagnosed with localized or metastatic breast cancer at the Paris Saint-Joseph Hospital Group (GhPSJ).
* Patients in whom adjuvant or neoadjuvant chemotherapy treatment is planned
* Patient affiliated to the social security system or, failing that, to another health insurance system
* Patient who has given written consent.

Exclusion Criteria:

* Psychotic patients (paranoia, schizophrenia and manic-depressive psychosis)
* Patient suffering from pathological dissociations
* Deaf and hard of hearing
* Blind and severely visually impaired
* Patient suffering from wounds or infections in the head area
* Patient suffering from respiratory disorders
* Patient with a high level of claustrophobia
* Patient whose investigator determines that he or she cannot wear a virtual reality helmet
* Patient under guardianship or curatorship
* Patient deprived of liberty.
* Pregnant or breastfeeding patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate, in patients undergoing chemotherapy for the treatment of breast cancer, the impact of the use of hypnotherapy performed by a virtual reality tool on the anxiety felt just before the PAC procedure. | Day 7
  Difference between the 2 groups of patients in terms of the anxiety felt just before the PAC procedure, evaluated by the Spielberger's State Anxiety Scale (STAI form Y-A).
  This scale evaluates the feelings of apprehension, tension, nervousness and anxiety that the subject feels at the time of the anxiety-provoking or competitive situation.

SECONDARY OUTCOMES:
Evaluate in patients undergoing chemotherapy for the treatment of breast cancer the impact of the use of hypnotherapy performed by a virtual reality tool on the maximum pain and its duration felt by patients since the insertion of PAC. | Day 7
  Difference between the 2 groups of patients in terms of maximum pain and its duration felt by the patients since PAC insertion evaluated on an numerical scale 30 minutes after PAC insertion
Evaluate in patients undergoing chemotherapy for the treatment of breast cancer the impact of the use of hypnotherapy using a virtual reality tool on the incidence of chemotherapy associated adverse events. | Day 7
  Difference between the 2 groups of patients in terms of frequency of nausea, vomiting, fatigue and peripheral neuropathies after chemotherapy cures, reported on questionnaire QLQ-C30
Evaluate in patients undergoing chemotherapy for the treatment of breast cancer the impact of the use of hypnotherapy using a virtual reality tool on quality of life as measured by the QLC30 scale at the end of chemotherapy. | 1 year
  Difference between the 2 groups of patients in terms of the score of the "globalhealth" section of the QLQ-C30 questionnaire at the end of chemotherapy
Evaluate in patients undergoing chemotherapy for the treatment of breast cancer the impact of the use of hypnotherapy using a virtual reality tool on the quality of life measured on the QBR23 scale at the end of chemotherapy. | 1 year
  Difference between the 2 groups of patients in terms of the quality of life score from the QLQ-QBR23 questionnaire at the end of the chemotherapy
Evaluate the impact of the use of hypnotherapy on the immune system in patients undergoing chemotherapy for the treatment of breast cancer using a virtual reality tool. | Day 7 and 1 year
  Difference between the 2 groups of patients in terms of IgA level evolution

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie GARNIER-VIOUGEAT, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France